CLINICAL TRIAL: NCT02430402
Title: Effect of Rehabilitation of Young Patients With Rheumatic Diseases in a Warm Climate. A Pilot Randomised Controlled Trial
Brief Title: Rehabilitation of Young Patients With Rheumatic Diseases in a Warm Climate
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 013.5
Record Dates: First submitted 2015-04-22; First posted 2015-04-30 (Estimated); Last update posted 2020-03-20 (Actual); Status verified 2020-03

CONDITIONS: Rheumatic Diseases
Keywords: Climatotherapy
MeSH Terms: conditions — Rheumatic Diseases | interventions — Rehabilitation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Climate therapy (Experimental): Climate therapy consisting of 3 week stay at rehabilitation facility in Spain
  Interventions: Other: Rehabilitation in warm climate
- Usual care (No Intervention): Usual care provided as needed / agreed between patient and health care providers

INTERVENTIONS:
Other: Rehabilitation in warm climate
  Arms: Climate therapy

SUMMARY:
Young patients with rheumatic diseases have challenges different from older patients due to their life situation. It has been reported that they do not have the same benefit from age non-specific rehabilitation in warm climate. This trial will test the effect of a specially adapted version of a rehabilitation program delivered in Spain (warm climate) for Norwegian young adults aged 20-35 years.

ELIGIBILITY:
Inclusion Criteria:

* Inflammatory rheumatic disease
* Self reliant in daily life

Exclusion Criteria:

- conditions that might influence ability to fly to Spain and participate in rehabilitation in warm climate (Unstable heart disease, Serious lung disease, Chronic open ulcers, Serious mental health conditions, alcohol or drug addiction, Intolerant of sun and heat)

Ages: 20 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2015-05 (Actual); Primary Completion 2017-08 (Actual); Study Completion 2017-08 (Actual)

PRIMARY OUTCOMES:
Coping (Effective Consumer Scale (EC17) | 12 months
  Measured with Effective Consumer Scale (EC17)
30 second sit to stand test | 12 months

SECONDARY OUTCOMES:
EQ5D | 12 months
Numerical Rating Scales (NRS) fatigue question | 12 months
Hannover functional Scale | 12 months
Coop Wonca | 12 months
Hopkins Symptom Checklist | 12 months
Patient Specific Functional scale | 12 months
Numerical Rating Scales (NRS) pain question | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Aslak Steinsbekk, PhD, Principal Investigator — Norwegian University of Science and Technology
Locations (1):
- Institute for Social Medicine, Trondheim, Norway

REFERENCES:
- [Result] Nilssen IR, Koksvik HS, Gronning K, Steinsbekk A. Rehabilitation in warm climate for young adults with inflammatory arthritis: A 12-month randomized controlled trial. J Rehabil Med. 2020 Apr 14;52(4):jrm00040. doi: 10.2340/16501977-2666. PMID 32179929